CLINICAL TRIAL: NCT00111748
Title: UARK 2005-01, A Phase III Study of Velcade, Thalidomide, and Dexamethasone (VTD) With or Without Adriamycin® in Relapsed/Refractory Patients
Brief Title: UARK 2005-01 Study of Velcade, Thalidomide, and Dexamethasone (VTD) With or Without Adriamycin® in Relapsed/Refractory Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Arkansas (Other)
Responsible Party: Nathan Petty, University_of_Arkansas
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 29432
Record Dates: First submitted 2005-05-24; First posted 2005-05-25 (Estimated); Last update posted 2015-10-06 (Estimated); Status verified 2015-10

CONDITIONS: Multiple Myeloma
Keywords: Myeloma
MeSH Terms: conditions — Multiple Myeloma; Neoplasms, Plasma Cell | interventions — Bortezomib; Thalidomide; Dexamethasone

ARMS (2):
- 1 (Active Comparator): Stratification:
  1. CA13/hypodiploidy at diagnosis versus no CA13/hypoploidy at diagnosis
  2. Prior Velcade vs. No prior Velcade
  TREATMENT:VTD Velcade 1.0 mg/m2 Days 1,4, 8,11 Thalidomide 100 mg Daily qhs Dexamethasone 20 mg Days 1, 2, 4,5, 8, 9, 11, 12 Lovenox 40 mg Days 1-14 Every 21 days
  Interventions: Drug: Velcade, Thalidomide, Dexamethasone
- 2 (Active Comparator): Stratification:
  1. CA13/hypodiploidy at diagnosis versus no CA13/hypoploidy at diagnosis
  2. Prior Velcade vs. No prior Velcade
  TREATMENT:
  VATD Velcade 1.0 mg/m2 Days 1,4, 8,11 Thalidomide 100 mg Daily qhs Dexamethasone 20 mg Days 1, 2, 4,5, 8, 9, 11, 12 Adriamycin 2.5 mg/m2 Days 1-4 & Days 9-12 Lovenox 40 mg Days 1-14 Every 21 days
  Interventions: Drug: Velcade, Thalidomide, Dexamethasone

INTERVENTIONS:
Drug: Velcade, Thalidomide, Dexamethasone — Dosage and Administration Schedule Each cycle will consist of 3 weeks (21 days). AGENT DOSE ROUTE DAYS Velcade 1.0 mg/m2 IV 1, 4, 8, and 11 Thalidomide 100 mg PO Daily, hs Dexamethasone 20 mg PO Days 1, 2, 4,5, 8, 9, 11, 12 Lovenox 40 mg SQ Days 1-14
  This 21-day period will be considered one treatment cycle; Cycle 2 would commence on Day 22 (Cycle 2, Day 1). The next cycle of treatment may be delayed up to day 29 due to non-toxicity reasons. Patients may continue to receive treatment every 21 days, provided there is no evidence of disease progression or no unacceptable toxicity for a maximum of eight cycles. At the discretion of the treating physician, patients may be eligible to receive treatment at their local physician after completion of the 1st cycle. These patients will need to return to MIRT prior to every cycle for cycles 2-4, cycles 6 and 8, and final visit.

SUMMARY:
The main goal of this study is to evaluate the effectiveness of the combination of these drugs, and whether they can be given safely together.

DETAILED DESCRIPTION:
In this study, there will be two arms (or groups). One arm will receive Velcade, thalidomide, and dexamethasone (VTD), and the other arm will receive VTD with Adriamycin.

This study has the following specific goal:

To evaluate the efficacy and toxicity of two treatments in multiple myeloma patients, relapsing after at least one course of high-dose treatment and an autologous stem cell transplant, or after at least two lines of conventional chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients with relapsing multiple myeloma (MM)
* Patients must have adequate platelet count of > 20,000 x 10^9/L, independent of transfusions, unless it is due to massive myeloma infiltration.
* Anticipated life expectancy of at least 3 months
* Ejection fraction by echocardiogram (ECHO) or multiple gated acquisition (MUGA) scan performed within 60 days prior to registration; left ventricular ejection fraction (LVEF) > 40% by ECHO or MUGA.
* Female patients of child bearing age are required to have a negative pregnancy test as indicated in thalidomide safety guidelines
* Patients must have a performance status of 0-2 based on Southwest Oncology Group (SWOG) criteria. Patients with a poor performance status (3-4), based solely on bone pain, will be eligible.
* All patients must be informed of the investigational nature of this study and must have signed an institutional review board (IRB)-approved informed consent in accordance with institutional and federal guidelines.

Exclusion Criteria:

* Evidence of central nervous system (CNS) involvement
* Grade > 2 peripheral neuropathy
* Hypersensitivity to Velcade, boron, or mannitol
* Recent (< 6 months) myocardial infarction, cerebrovascular accident (CVA)/stroke, unstable angina, difficult to control congestive heart failure, uncontrolled hypertension, or difficult to control cardiac arrhythmias.
* Evidence of chronic obstructive or chronic restrictive pulmonary disease.
* Prior malignancy, except for adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, or other cancer for which the patient has been disease free for at least three years.
* Patients must not have significant co-morbid medical conditions or uncontrolled life threatening infection.
* Pregnant or nursing women. Women of child-bearing potential must have a negative pregnancy test documented within one week of registration. Women and men of reproductive potential may not participate unless they have agreed to use an effective contraceptive method for the duration of the study treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2005-02; Primary Completion 2006-09 (Actual); Study Completion 2006-09 (Actual)

PRIMARY OUTCOMES:
Evaluate the effectiveness of the combination of these drugs | 168 days

SECONDARY OUTCOMES:
Evaluate the efficacy and toxicity of two treatments in multiple myeloma patients, relapsing after at least one course of high-dose treatment and an autologous stem cell transplant | 168 days

CONTACTS AND LOCATIONS:
Overall Officials: Klaus Hollmig, MD, Principal Investigator — University of Arkansas
Locations (1):
- University of Arkansas for Medical sciences, Little Rock, Arkansas, United States